CLINICAL TRIAL: NCT03242642
Title: Transcatheter Mitral Valve Replacement With the Medtronic Intrepid™ TMVR System in Patients With Severe Symptomatic Mitral Regurgitation - APOLLO Trial
Brief Title: Transcatheter Mitral Valve Replacement With the Medtronic Intrepid™ TMVR System in Patients With Severe Symptomatic Mitral Regurgitation.
Acronym: APOLLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17022TMV001
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Mitral Valve Regurgitation
Keywords: Heart disease; valve disease; heart valve disease; mitral regurgitation; cardiovascular disease; mitral insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Diseases; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Primary Cohort- TMVR (Experimental): Treatment of mitral regurgitation with the Medtronic Transcatheter Mitral Valve Replacement System (TMVR)
  Interventions: Device: Medtronic Intrepid Transcatheter Mitral Valve Replacement System (TMVR)
- Mitral Annular Calcification -TMVR (Experimental): Treatment of mitral regurgitation with the Medtronic Transcatheter Mitral Valve Replacement System (TMVR)
  Interventions: Device: Medtronic Intrepid Transcatheter Mitral Valve Replacement System (TMVR)

INTERVENTIONS:
Device: Medtronic Intrepid Transcatheter Mitral Valve Replacement System (TMVR) — mitral valve replacement
Device: Medtronic Intrepid Transcatheter Mitral Valve Replacement System (TMVR) — Medtronic Intrepid Transcatheter Mitral Valve Replacement System (TMVR) mitral valve replacement

SUMMARY:
Multi-center, global, prospective, non-randomized, interventional, pre-market trial. All subjects enrolled with receive the study device.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe or severe symptomatic mitral regurgitation
* Local site multidisciplinary heart team experienced in mitral valve therapies agrees that the subject is unsuitable for treatment with approved transcatheter repair or conventional mitral valve intervention

Exclusion Criteria:

* prior transcatheter mitral valve procedure with device currently implanted
* anatomic contraindications
* prohibitive mitral annular calcification
* left ventricular ejection fraction <25%
* need for emergent or urgent surgery
* hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2036-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Cohort | 1 year
  Composite of all-cause mortality or heart failure hospitalization
MAC Cohort | 1 year
  All-cause mortality

SECONDARY OUTCOMES:
All-cause mortality, disabling stroke, acute kidney injury, prolonged ventilation, deep wound infection, reoperation or reintervention, and major bleeding | 30 days or hospital discharge (whichever is later)
  Composite
Degree of mitral regurgitation | 6 months
  measured by echocardiography
Quality of Life Improvement | 3 months (KCCQ)
  measured by KCCQ
Change in New York Heart Association Class | 30 days
  change in NYHA Class
Echocardiographic assessments of degree mitral valve regurgitation | 1 year
  measured by echocardiography
Cardiovascular hospitalizations | 1 year
  cardiovascular hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mack, MD, Study Chair — Baylor Scott & White Hospital; David Adams, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Martin Leon, MD, Principal Investigator — New York Presbyterian Hospital/Columbia University Medical Center
Locations (85):
- United States (78):
  - University of Alabama Birmingham (UAB) Hospital, Birmingham, Alabama
  - Abrazo Heart Hospital, Phoenix, Arizona
  - Scripps Memorial Hospital, La Jolla, California
  - PIH Health Good Samaritan Hospital, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Keck Hospital of the University of Southern California, USC, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - Morton Plant, Clearwater, Florida
  - HealthPark Medical Center, Fort Myers, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - MercyOne Des Moines Medical Center, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Saint John Hospital, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center - East Bank, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Providence St Patrick, Missoula, Montana
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Northwell Health North Shore University Hospital, Manhasset, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - New York-Presbyterian Hospital Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - Saint Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health & Science University Hospital, Portland, Oregon
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - CHI Saint Luke's Health-Baylor Saint Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Hospital, San Antonio, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Saint Mary's Hospital/Bon Secours, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - The Swedish Medical Center Cherry Hill, Seattle, Washington
  - University of Washington (UW) Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (6):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Saint Paul's Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Montreal Heart Insitute, Montreal, Quebec
  - Glen Royal Victoria Hospital, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Tang GHL, Rajagopal V, Sorajja P, Bajwa T, Gooley R, Walton A, Modine T, Ng MK, Williams MR, Zajarias A, Hildick-Smith D, Tchetche D, Spargias K, Rajani R, Bapat VN, De Backer O, Blackman D, McCarthy P, Laine M, Jain R, Martin R, Thaden JJ, Marka NA, Mack M, Adams DH, Leon MB, Reardon MJ. Five-year outcomes of the early-generation Intrepid transapical transcatheter mitral valve replacement system. EuroIntervention. 2026 Feb 2;22(3):e172-e182. doi: 10.4244/EIJ-D-25-01133. PMID 41251714